CLINICAL TRIAL: NCT07299097
Title: Epidemiology of Narcolepsy Type 1 and Type 2 in Spain
Acronym: HYPNOS
Status: Not yet recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-861-4006
Record Dates: First submitted 2025-12-10; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Narcolepsy Type 1; Narcolepsy Type 2
Keywords: Drug therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Core Group: Participants with Narcolepsy Type (NT1) and Narcolepsy Type (NT2) of any age, ethnicity and nationality, treated / under follow-up in approximately 10 Spanish public hospitals, who are alive at any point during 2023 or 2024, residing in the hospitals' reference areas will be retrospectively observed through chart reviews. The retrospective data for up to approximately 10 years would be assessed.
  Interventions: Other: No intervention
- Supplementary Group: Participants with NT1 and NT2 from Spain will undergo an online survey conducted in collaboration with a patient advocacy group.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — As this is an observational study, no intervention will be administered.

SUMMARY:
The main purpose of this study is to find out how many people in Spain have been diagnosed with narcolepsy type 1 and type 2, and how many new participants are diagnosed each year. Narcolepsy is a rare sleep disorder that causes excessive daytime sleepiness. The researchers will look at medical records from hospitals across Spain to count participants with these conditions and understand patterns in diagnosis over time.

DETAILED DESCRIPTION:
The aim is to do epidemiology study in the core group thus the enrolment number is not applicable to this group, however approximately100 participants in the supplementary group (online survey).

ELIGIBILITY:
- Core Group:

Inclusion Criteria:

1. Participants with NT1 or NT2 following International Classification of Sleep Disorders, 3rd Edition (ICSD-3) or ICSD-3 text revision (ICSD-3-TR) criteria who are alive at any point during 2023 or 2024.
2. Any age, ethnicity and nationality.
3. Treated / under follow-up in the study site and residing in the hospitals' reference areas. Consideration will be given if participants have changed their address or reached adulthood.

Exclusion Criteria

1. NT1 or NT2 participants who do not reside in the hospitals' reference areas.

- Supplementary Group:

Inclusion criteria:

1. Confirmation to have a diagnosis of NT1 or NT2 by a specialist.
2. Participants greater than equal to (≥) 18 years or parents of narcolepsy participants under 18 years of age.
3. Any gender, ethnicity or nationality.
4. Residence in Spain.

Exclusion criteria:

1. Participants without a confirmed NT1 or NT2 diagnosis by a specialist.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with NT1 and NT2 from Spain.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Core Group: Prevalence of Participants With NT1 and NT2 per 100,000 Population | Up to 1 year
  The overall study prevalence will be calculated as the number of participants diagnosed with NT1 and NT2 from all public hospitals reporting cases divided by number of people living in the areas served by these hospitals resulting in a study prevalence fraction. The study prevalence fraction will be then extrapolated to the Spanish population to estimate the standardized overall prevalence of NT1 and NT2 in Spain.
Core Group: Prevalence of Adult Participants With NT1 and NT2 per 100,000 Adult Population | Up to 1 year
  The overall study prevalence will be calculated as the number of adult participants diagnosed with NT1 and NT2 from all public hospitals reporting cases divided by number of adult people living in the areas served by these hospitals resulting in a study prevalence fraction. The study prevalence fraction will be then extrapolated to the Spanish population to estimate the standardized overall prevalence of NT1 and NT2 in Spain.
Core Group: Prevalence of Paediatric/Adolescent Participants With NT1 and NT2 per 100,000 Paediatric/Adolescent Population | Up to 1 year
  The overall study prevalence will be calculated as number of diagnosed paediatric/adolescent participants from all public hospitals divided by number of paediatric/adolescent living in the areas served by these hospitals resulting in a study prevalence fraction. The study prevalence fraction will be then extrapolated to the Spanish population to estimate the standardized overall prevalence of NT1 and NT2 in Spain.
Core Group: Prevalence of Male Participants With NT1 and NT2 per 100,000 Male Population | Up to 1 year
  The overall study prevalence will be calculated as the number of male participants diagnosed with NT1 and NT2 from all public hospitals reporting cases divided by number of males living in the areas served by these hospitals resulting in a study prevalence fraction. The study prevalence fraction will be then extrapolated to the Spanish population to estimate the standardized overall prevalence of NT1 and NT2 in Spain.
Core Group: Prevalence of Female Participants With NT1 and NT2 per 100,000 Females Population | Up to 1 year
  The overall study prevalence will be calculated as the number of female participants diagnosed with NT1 and NT2 from all public hospitals reporting cases divided by number of females living in the areas served by these hospitals resulting in a study prevalence fraction. The study prevalence fraction will be then extrapolated to the Spanish population to estimate the standardized overall prevalence of NT1 and NT2 in Spain.
Core Group: Incidence of NT1 and NT2 per 100,000 Population | Up to 2 years
  The incidence for both the years will be calculated as (average of both years). And for each year, the number of participants diagnosed for the first time from all hospitals divided by number of people living in the areas served by the hospitals resulting in a study incidence fraction. The study incidence fraction will be then extrapolated to the Spanish population to estimate the standardized overall incidence of NT1 and NT2 in Spain.
Core Group: Incidence of NT1 and NT2 per 100,000 Adult Population | Up to 2 years
  The incidence for both the years will be calculated as (average of both years) and for each year, the number of adult participants diagnosed for the first time from all hospitals divided by number of adults living in the areas served by these hospitals resulting in a study incidence fraction. The study incidence fraction will be then extrapolated to the Spanish population to estimate the standardized overall incidence of NT1 and NT2 in Spain.
Core Group: Incidence of Paediatric/Adolescent NT1 and NT2 per 100,000 Paediatric/Adolescent Population | Up to 2 years
  The incidence for both the years will be calculated as (average of both years) and for each year, the number of paediatric/adolescent participants diagnosed for the first time from all hospitals divided by number of paediatric/adolescent living in the areas served by these hospitals resulting in a study incidence fraction. The study incidence fraction will be then extrapolated to the Spanish population to estimate the standardized overall incidence of NT1 and NT2 in Spain.
Core Group: Incidence of Male NT1 and NT2 per 100,000 Male Population | Up to 2 years
  The incidence for both the years will be calculated as (average of both years) and for each year, the number of male participants diagnosed for the first time from all hospitals divided by number of male participants living in the areas served by these hospitals resulting in a study incidence fraction. The study incidence fraction will be then extrapolated to the Spanish population to estimate the standardized overall incidence of NT1 and NT2 in Spain.
Core Group: Incidence of Female NT1 and NT2 per 100,000 Female Population | Up to 2 years
  The incidence for both the years will be calculated as (average of both years) and for each year, the number of female participants diagnosed for the first time from all hospitals divided by number of female participants living in the areas served by these hospitals resulting in a study incidence fraction. The study incidence fraction will be then extrapolated to the Spanish population to estimate the standardized overall incidence of NT1 and NT2 in Spain.
Supplementary Group: Number of Participants with NT1 and NT2 who Attend Regular Follow-ups | On a day of survey (any 1 day) during the study for each participant
  Proportion of Participants with NT1 and NT2 in Spain who attended regular follow ups at only public hospitals, only private hospitals, and both private and public hospitals will be reported.

SECONDARY OUTCOMES:
Core Group: Proportion of Participants as per Gender with NT1 and NT2 at Diagnosis | Up to approximately 10 years
Core Group: Proportion of Participants as per Age with NT1 and NT2 at Diagnosis | Up to approximately 10 years
Core Group: Proportion of Participants as per Gender with NT1 and NT2 at Symptom Onset | Up to approximately 10 years
Core Group: Proportion of Participants as per Age with NT1 and NT2 at Symptom Onset | Up to approximately 10 years
Core Group: Percentage Change in NT1 and NT2 Prevalence Over Past 10 Years | Up to 10 years
  The overall prevalence will be calculated as the number of participants diagnosed with NT1 and NT2 from all public hospitals reporting cases divided by number of people living in the areas served by these hospitals resulting in prevalence fraction. The overall percentage change of participant resulting from the above method will be reported.
Core Group: Percentage Change in Adult With NT1 and NT2 Prevalence Over Past 10 Years | Up to 10 years
  The overall prevalence will be calculated as the number of adult participants diagnosed with NT1 and NT2 from all public hospitals reporting cases divided by number of adult people living in the areas served by these hospitals resulting in a study prevalence fraction. The overall percentage change of participant resulting from the above method will be reported.
Core Group: Percentage Change in Paediatric/Adolescent NT1 and NT2 Prevalence Over Past 10 Years | Up to 10 years
  The overall prevalence will be calculated as the number of paediatric/adolescent participants diagnosed with NT1 and NT2 from all public hospitals reporting cases divided by number of paediatric/adolescent living in the areas served by these hospitals resulting in a study prevalence fraction. The overall percentage of participant resulting from the above method will be reported.
Core Group: Percentage Change in NT1 and NT2 Incidence Over Past 10 Years | Up to 10 years
  The incidence will be calculated as number of participants diagnosed for the first time from all hospitals divided by number of people living in the areas served by these hospitals resulting in a study incidence fraction. The overall percentage change of participant resulting from the above method will be reported.
Core Group: Percentage Change in Adult NT1 and NT2 Incidence Over Past 10 Years | Up to 10 years
  The incidence will be calculated as number of adult participants diagnosed for the first time from all hospitals divided by number of adults living in the areas served by these hospitals resulting in a study incidence fraction. The overall percentage change of participant resulting from the above method will be reported.
Core Group: Percentage Change in Paediatric/Adolescent NT1 and NT2 Incidence Over Past 10 Years | Up to 10 years
  The incidence will be calculated as number of paediatric/adolescent participants diagnosed for the first time from all hospitals divided by number of paediatric/adolescent living in the areas served by these hospitals resulting in a study incidence fraction. The overall percentage of participant resulting from the above method will be reported.
Core Group: Diagnostic Delay for Incident Participants with NT1 and NT2 | Up to approximately 10 years
  Diagnostic delay means that cases that began to present symptoms in the years prior to one year and have not yet been diagnosed.
Core Group: Diagnostic Delay for Incident Adult Participants with NT1 and NT2 | Up to approximately 10 years
  Diagnostic delay means that cases that began to present symptoms in the years prior to one year and have not yet been diagnosed.
Core Group: Diagnostic Delay for Incident Paediatric/Adolescent Participants with NT1 and NT2 | Up to approximately 10 years
  Diagnostic delay means that cases that began to present symptoms in the years prior to one year and have not yet been diagnosed.
Core Group: Diagnostic Delay for Incident Male Participants with NT1 and NT2 | Up to approximately 10 years
  Diagnostic delay means that cases that began to present symptoms in the years prior to one year and have not yet been diagnosed.
Core Group: Diagnostic Delay for Incident Female Participants with NT1 and NT2 | Up to approximately 10 years
  Diagnostic delay means that cases that began to present symptoms in the years prior to one year and have not yet been diagnosed.
Core Group: Percentage Change in Diagnostic Delay for Participants With NT1 and NT2 Over Past 10 Years | Up to 10 years
Core Group: Percentage Change in Diagnostic Delay for Adult Participants With NT1 and NT2 Over Past 10 Years | Up to 10 years
Core Group: Percentage Change in Diagnostic Delay for Paediatric/Adolescent Participants With NT1 and NT2 Over Past 10 Years | Up to 10 years
Core Group: Percentage Change in Diagnostic Delay for Male Participants With NT1 and NT2 Over Past 10 Years | Up to 10 years
Core Group: Percentage Change in Diagnostic Delay for Female Participants With NT1 and NT2 Over Past 10 Years | Up to 10 years
Supplementary Group: Proportion of Participants With NT1 and NT2 who Were Diagnosed at Public hospitals and Private Practices | On a day of survey (any 1 day) during the study for each participant
Supplementary Group: Proportion of Participants who Choose to be Followed in Public, Private, or Both Types of Hospitals and Reasons | On a day of survey (any 1 day) during the study for each participant
Supplementary Study: Age at symptom onset | On a day of survey (any 1 day) during the study for each participant
Supplementary Study: Age at diagnosis | On a day of survey (any 1 day) during the study for each participant
Supplementary Study: Proportion of Participants as per Speciality of the Doctor Visited First for Narcolepsy Symptoms | On a day of survey (any 1 day) during the study for each participant
Supplementary Study: Proportion of Participants as per Speciality of the Doctor who Diagnosed Narcolepsy | On a day of survey (any 1 day) during the study for each participant
Supplementary Study: Number of Doctors Visited by Participant Prior to Receiving a Narcolepsy Diagnosis | On a day of survey (any 1 day) during the study for each participant
Supplementary Study: Proportion of Participants With Misdiagnosis Prior to Narcolepsy Diagnosis | On a day of survey (any 1 day) during the study for each participant
Supplementary Study: Proportion of Participants with Comorbidities | On a day of survey (any 1 day) during the study for each participant
Supplementary Study: Proportion of Participants as per Place of Residence (Autonomous Community) | On a day of survey (any 1 day) during the study for each participant

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/